CLINICAL TRIAL: NCT06135467
Title: Association Between MAFLD ( Metabolic Associated Fatty Liver Disease) and Chronic Kidney Disease
Brief Title: Association Betweenq MAFLD ( Metabolic Associated Fatty Liver Disease) and Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa adel shehata, Doctor, Assiut University
Other Study IDs: Mafld in ckd patients
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Mafld in Ckd Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess frequency of renal affection in mafld

DETAILED DESCRIPTION:
Metabolic dysfunction-associated fatty liver disease (MAFLD) is a multisystem disorder, but its relationship with kidney injury remains controversial. This study aimed to evaluate MAFLD effects on the chronic kidney disease (CKD) frequency The association between metabolic dysfunction associated fatty liver disease (MAFlD) and extrahepatic disease is not known .the aim of this cross sectional study is to compare the frequency of CKD in patients with MAFLD and examine association between presence and severity of MAFLD and CKD and abnormal albuminuria.

Non-alcoholic fatty liver disease (NAFLD) is characterized by the accumulation of fat in more than 5% of hepatocytes in the absence of excessive alcohol consumption and other secondary causes of hepatic steatosis. In 2020, the more inclusive term metabolic (dysfunction)-associated fatty liver disease (MAFLD) - defined by broader diagnostic criteria - was proposed to replace the term NAFLD. The new terminology and revised definition better emphasize the pathogenic role of metabolic dysfunction and uses a set of definitive, inclusive criteria for diagnosis. Diagnosis of MAFLD is based on evidence of hepatic steatosis (as assessed by liver biopsy, imaging techniques or blood biomarkers and scores) in persons who are overweight or obese and have type 2 diabetes mellitus or metabolic dysregulation, regardless of the coexistence of other liver diseases or excessive alcohol consumption.

The known association between NAFLD and chronic kidney disease (CKD) and our understanding that CKD can occur as a consequence of metabolic dysfunction suggests that individuals with MAFLD - who by definition have fatty liver and metabolic comorbidities - are at increased risk of CKD.

MAFLD appears to be tightly linked to incident chronic kidney disease (CKD). This association may be attributed to multiple shared risk factors including type 2 diabetes mellitus, arterial hypertension, obesity, dyslipidemia, and insulin resistance Diagnostic criteria of MAFLD are ( steatosis with one of the following

1. BMI >25
2. type II DM
3. > 2 metabolic abnormalities [ 1)waist circumferance >94 in males or 80 in females 2)bp >130/85 3) plasma triglycrides > 150 mg / dl 4) HDL < 40 5)prediabetes 6) HOMA insulin resistance score >2.5 7)plasma hs CRP> 2 mg/dl ]

ELIGIBILITY:
Inclusion Criteria:

1. CKD patients type II . III and type IV not on dialysis
2. Patients with MAFLD
3. patients with type II DM

Exclusion Criteria:

1. Patients with AKI
2. patients with NAFLD
3. patients with alcoholic fatty liver disease
4. patients with type I DM
5. malignancy
6. HBV HCV
7. autoimmune disease
8. liver cirrhosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study is done on 150 patients diagnosed as MAFLD with its diagnostic criteria (Diagnostic criteria of MAFLD are ( steatosis with one of the following
  1. BMI >25
  2. type II DM
  3. > 2 metabolic abnormalities [ 1)waist circumferance >94 in males or 80 in females 2)bp >130/85 3) plasma triglycrides > 150 mg / dl 4) HDL < 40 5)prediabetes 6) HOMA insulin resistance score >2.5 7)plasma hs CRP> 2 mg/dl ].
  And divided into 3 groups :
  1. MAFLD with type II DM
  2. MAFLD not type II DM
  3. control group
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
the frequency of MAFLD in CKD patients 2_To screen early MAFLD in CKD patients 3_To association between MAFLD in CKD and type II DM patients | Baseline
  estimate the frequency of MAFLD in CKD patients 2_To screen early MAFLD in CKD patients 3_To association between MAFLD in CKD and type II DM patients